CLINICAL TRIAL: NCT02348658
Title: A Phase 1, Randomized, Open-Label, Crossover Study to Evaluate the Food-Effect of Single Oral Dose of TAK-536TCH Final Formulation Tablet in Healthy Adult Male Subjects
Brief Title: A Phase 1 Food Effect Study of TAK-536TCH Final Formulation Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TAK-536TCH/CPH-004; U1111-1165-5595 (Registry Identifier: WHO); JapicCTI-152777 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-01-15; First posted 2015-01-28 (Estimated); Results first posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-03

CONDITIONS: Hypertension
Keywords: Pharmacological therapy
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasted dosing followed by fed dosing (Other): Dosing in the fasted state followed by fed dosing
  Interventions: Drug: TAK-536TCH
- Fed dosing followed by fasted dosing (Other): Dosing in the fed state followed by fasted dosing
  Interventions: Drug: TAK-536TCH

INTERVENTIONS:
Drug: TAK-536TCH — TAK-536TCH tablets

SUMMARY:
This is a phase 1, randomized, open-label, crossover study to evaluate the food-effect of single oral dose of TAK-536TCH final formulation tablet in healthy adult male participants.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the food effect on the pharmacokinetics and safety of a single oral dose of TAK-536TCH under fasted and fed conditions in the morning in healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria:

* 1. In the opinion of the investigator and subinvestigator, the participant is capable of understanding and complying with protocol requirements.

  2. The participant signs and dates a written, informed consent form prior to the initiation of any study procedures.

  3. The participant is a healthy Japanese adult male. 4. The participant is aged 20 to 35 years, inclusive at the time of informed consent.

  5. The participant weighs at least 50.0 kg and has a body mass index (BMI) from 18.5 to 25.0 kilograms per square meter (kg/m^2), inclusive at Screening.

Exclusion Criteria:

1. Participant has systolic blood pressure less-than (<) 90 millimeters of mercury (mmHg) at Screening.
2. Participant has suspected hypotension and associated physical findings, such as dizziness postural, facial pallor, or cold sweats based on evaluation/physical examination at Screening, on Day -1 of Period 1, or up to administration on the Period 1.
3. The participant has received any study drug within 16 weeks (that is [i.e.], 112 days) prior to study drug administration of Period 1.
4. The participant has received TAK-491*, TAK-536, amlodipine, or hydrochlorothiazide in a previous clinical study or as a therapeutic agent.
5. The participant has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urological, or endocrine disease, or other abnormality (other than the disease studied), which could impact the ability of the participant to participate or potentially confound the study results.
6. Participant has a known hypersensitivity to drugs.
7. Participant has a positive urine drug result for drugs of abuse at Screening.
8. Participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 2 years prior to the Screening visit or was unwilling to agree to abstain from alcohol and drugs throughout the study.
9. Participant required any prohibited concomitant drugs, vitamins, or food products listed in the prohibited concomitant drugs and foods table.
10. Participant has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (i.e., a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn, or any surgical intervention [e.g., cholecystectomy]).
11. Participant has a history of cancer.
12. Participant has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody/antigen, or serological reactions for syphilis at Screening.
13. Participant has poor peripheral venous access.
14. Participant has undergone whole blood collection of at least 200 mL within 4 weeks (28 days) or at least 400 mL within 12 weeks (84 days) prior to study drug administration in Period 1.
15. Participant has undergone whole blood collection of at least 800 mL in total within 52 weeks (364 days) prior to study drug administration in Period 1.
16. Participant has undergone blood component collection within 2 weeks (14 days) prior to study drug administration in Period 1.
17. Participant has a hemoglobin value of less than 12.5 g/dL in laboratory testing at Screening or prior to study drug administration in Period 1.
18. Participant has a clinically significant ECG abnormality at Screening or prior to study drug administration in Period 1.
19. Participant has abnormal laboratory values at Screening or prior to study drug administration of Period 1 that suggest a clinically significant underlying disease or participant with the following lab abnormalities: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is >1.5-fold the upper limits of normal range.
20. Participant who, in the opinion of the investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Manager, Study Chair — Takeda
Locations (1):
- Fukuoka, Fukuoka, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 29 January 2015 to 11 March 2015.
Pre-assignment Details: Healthy adult male participants were enrolled in 1 of 2 treatment sequences in either of the Periods 1 or 2: Sequence A: TAK-536TCH (combination drug of TAK-536 [azilsartan], amlodipine besilate [AML], hydrochlorothiazide [HTZ]) Fasted in Period 1+ TAK-536TCH Fed in period 2; Sequence B: TAK-536TCH Fed in Period 1+ TAK-536TCH Fasted in Period 2.
Groups:
- TAK-536TCH Fasted + TAK-536TCH Fed: TAK-536TCH (20 milligram [mg]/5 mg/12.5 mg), tablet, in fasted condition, orally, once on Day 1 in Period 1, followed by 22 days washout period, followed by TAK-536TCH (20 mg/5 mg/12.5 mg), tablet, in fed condition, orally, once on Day 1 in Period 2.
- TAK-536TCH Fed + TAK-536TCH Fasted: TAK-536TCH (20 mg/5 mg/12.5 mg), tablet, in fed condition, orally, once on Day 1 in Period 1, followed by 22 days washout period, followed by TAK-536TCH (20 mg/5 mg/12.5 mg), tablet, in fasted condition, orally, once on Day 1 in Period 2.
Period: Period 1 (7 Days)
Arm/Group | TAK-536TCH Fasted + TAK-536TCH Fed | TAK-536TCH Fed + TAK-536TCH Fasted
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout Period (22 Days)
Arm/Group | TAK-536TCH Fasted + TAK-536TCH Fed | TAK-536TCH Fed + TAK-536TCH Fasted
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Period 2 (7 Days)
Arm/Group | TAK-536TCH Fasted + TAK-536TCH Fed | TAK-536TCH Fed + TAK-536TCH Fasted
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pharmacokinetic (PK) analysis set included all participants who received the study drug, completed the minimum protocol-specified procedures without any major protocol deviations, and who were evaluable for the food-effect.
Groups:
- All Participants: All participants who received either 1 of the two treatment sequences: Sequence 1: TAK-536TCH (20 mg/5 mg/12.5 mg), tablet, in fasted condition, orally, once on Day 1 in Period 1, followed by 22 days washout period, followed by TAK-536TCH (20 mg/5 mg/12.5 mg), tablet, in fed condition, orally, once on Day 1 in Period 2 or Sequence 2: TAK-536TCH (20 mg/5 mg/12.5 mg), tablet, in fed condition, orally, once on Day 1 in Period 1, followed by 22 days washout period, followed by TAK-536TCH (20 mg/5 mg/12.5 mg), tablet, in fasted condition, orally, once on Day 1 in Period 2.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.2 (3.54)
Sex/Gender, Customized [Number; unit: participants]
  Male | 12
Region of Enrollment [Number; unit: participants]
  Japan | 12
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 171.3 (6.03)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 61.18 (5.548)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 20.85 (1.499)
Smoking Classification [Number; unit: participants]
  Never Smoked | 6
  Current Smoker | 3
  Ex-Smoker | 3
Alcohol Classification [Number; unit: participants]
  Drinks a few Days per Month | 7
  Had Never Drunk | 5
Caffeine Classification [Number; unit: participants]
  Caffeine Consumer | 1
  Caffeine Non-Consumer | 11

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Plasma Concentration for TAK-536, Its Metabolites (M-I and M-II) and Hydrochlorothiazide (HCTZ)
Time Frame: Day 1: predose and at multiple time points (up to 48 hours) postdose in each period
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- TAK-536TCH Fasted: TAK-536TCH (20 mg/5 mg/12.5 mg), tablet, in fasted condition, orally, once on Day 1 in either Period 1 or Period 2.
- TAK-536TCH Fed: TAK-536TCH (20 mg/5 mg/12.5 mg), tablet, in fed condition, orally, once on Day 1 in either Period 1 or Period 2.
Arm/Group | TAK-536TCH Fasted | TAK-536TCH Fed
Number analyzed (Participants) | 12 | 12
nanogram per milliliter (ng/mL)
  TAK-536 | 1912.0 (253.39) | 1783.7 (318.16)
  M-I | 448.3 (143.36) | 455.3 (131.68)
  M-II | 453.5 (109.75) | 451.9 (101.18)
  HCTZ | 119.4 (30.481) | 101.6 (14.700)

2. Primary Outcome: Cmax: Maximum Plasma Concentration for Amlodipine Besilate (AML)
Time Frame: Day 1: predose and at multiple time points (up to 120 hours) postdose in each period
Population: PK analysis set included all participants who received the study drug, completed the minimum protocol-specified procedures without any major protocol deviations, and who were evaluable for the food-effect.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-536TCH Fasted | TAK-536TCH Fed
Number analyzed (Participants) | 12 | 12
ng/mL | 3.752 (0.5124) | 3.668 (0.6468)

3. Primary Outcome: AUC(0-48): Area Under the Plasma Concentration-Time Curve From Time 0 to 48 Hours Postdose in Each Period for TAK-536, Its Metabolites (M-I and M-II) and HCTZ
Description: AUC(0-48) is a measure of the area under the plasma concentration time-curve from time 0 to 48 hours postdose.
Time Frame: Day 1: predose and at multiple time points (up to 48 hours) postdose in each period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | TAK-536TCH Fasted | TAK-536TCH Fed
Number analyzed (Participants) | 12 | 12
nanogram*hour per milliliter (ng*hr/mL)
  TAK-536 | 14599.8 (2254.31) | 13279.4 (2889.22)
  M-I | 3215.8 (698.75) | 2693.8 (706.41)
  M-II | 9093.3 (1711.69) | 8990.8 (2310.99)
  HCTZ | 670.8 (75.912) | 595.2 (68.915)

4. Primary Outcome: AUC(0-120): Area Under the Plasma Concentration-Time Curve From Time 0 to 120 Hours Postdose in Each Period for AML
Description: AUC(0-120) is a measure of the area under the plasma concentration time-curve from time 0 to 120 hours postdose.
Time Frame: Day 1: predose and at multiple time points (up to 120 hours) postdose in each period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-536TCH Fasted | TAK-536TCH Fed
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 119.370 (27.7395) | 125.749 (26.9893)

5. Primary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration in Each Period for TAK-536, Its Metabolites (M-I and M-II) and HCTZ
Description: AUC(0-tlqc) is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (AUC[0-tlqc]).
Time Frame: Day 1: predose and at multiple time points (up to 48 hours) postdose in each period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-536TCH Fasted | TAK-536TCH Fed
Number analyzed (Participants) | 12 | 12
ng*hr/mL
  TAK-536 | 14599.8 (2254.31) | 13279.4 (2889.22)
  M-I | 3215.8 (698.75) | 2693.8 (706.41)
  M-II | 9093.3 (1711.69) | 8990.8 (2310.99)
  HCTZ | 641.3 (87.752) | 556.4 (70.514)

6. Primary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration in Each Period for AML
Description: as for outcome 5
Time Frame: Day 1: predose and at multiple time points (up to 120 hours) postdose in each period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-536TCH Fasted | TAK-536TCH Fed
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 119.370 (27.7395) | 125.749 (26.9893)

7. Primary Outcome: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity in Each Period for TAK-536, Its Metabolites (M-I and M-II) and HCTZ
Description: AUC (0-inf) is a measure of total plasma exposure to the drug from time zero extrapolated to infinity.
Time Frame: Day 1: predose and at multiple time points (up to 48 hours) postdose in each period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-536TCH Fasted | TAK-536TCH Fed
Number analyzed (Participants) | 12 | 12
ng*hr/mL
  TAK-536 | 15077.4 (2433.01) | 13700.9 (3154.23)
  M-I | 3271.3 (708.48) | 2755.1 (727.37)
  M-II | 10496.0 (2221.49) | 10193.0 (2804.33)
  HCTZ | 673.5 (87.075) | 595.9 (69.847)

8. Primary Outcome: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for AML
Description: AUC (0-inf) is a measure of total plasma exposure to the drug from time zero extrapolated to infinity.
Time Frame: Day 1: predose and at multiple time points (up to 120 hours) postdose in each period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-536TCH Fasted | TAK-536TCH Fed
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 132.941 (37.5121) | 140.484 (34.4402)

9. Primary Outcome: Urinary Excretion Ratio of TAK-536, Its Metabolites (M-I and M-II) and HCTZ
Description: Urinary excretion ratio (percent [%] of dose) of TAK-536, its metabolite M-I, M-II and HCTZ in urine were calculated for each participant. Ratio was calculated from the urine concentrations of each analyte and the volume of urine collected in each pooling period.
Time Frame: Day 1: predose and at multiple time-points (up to 48 hours) postdose in each period
Population: as for outcome 2
Measure: Number; unit: percentage of dose
Arm/Group | TAK-536TCH Fasted | TAK-536TCH Fed
Number analyzed (Participants) | 12 | 12
percentage of dose
  TAK-536 | 13.682 | 13.080
  M-I | 0.076 | 0.033
  M-II | 19.275 | 19.933
  HCTZ | 73.742 | 74.042

10. Primary Outcome: Urinary Excretion Ratio of AML
Description: Urinary excretion ratio (% of dose) of AML in urine were calculated for each participant. Ratio was calculated from the urine concentrations of each analyte and the volume of urine collected in each pooling period.
Time Frame: Day 1: predose and at multiple time-points (up to 120 hours) postdose in each period
Population: as for outcome 2
Measure: Number; unit: percentage of dose
Arm/Group | TAK-536TCH Fasted | TAK-536TCH Fed
Number analyzed (Participants) | 12 | 12
percentage of dose | 6.843 | 7.328

11. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Time Frame: Baseline up to 14 days after last dose of study drug (14 days after Day 1 of Period 2 )
Population: Safety analysis set included all participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | TAK-536TCH Fasted | TAK-536TCH Fed
Number analyzed (Participants) | 12 | 12
participants | 1 | 1

12. Secondary Outcome: Number of Participants With TEAEs Related to Vital Signs
Time Frame: Baseline up to 14 days after last dose of study drug (14 days after Day 1 of Period 2 )
Population: Safety analysis set included all participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | TAK-536TCH Fasted | TAK-536TCH Fed
Number analyzed (Participants) | 12 | 12
participants | 0 | 0

13. Secondary Outcome: Number of Participants With TEAEs Related to Body Weight
Time Frame: Baseline up to 14 days after last dose of study drug (14 days after Day 1 of Period 2 )
Population: Safety analysis set included all participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | TAK-536TCH Fasted | TAK-536TCH Fed
Number analyzed (Participants) | 12 | 12
participants | 0 | 0

14. Secondary Outcome: Number of Participants With TEAEs Categorized Into Investigations System Organ Class (SOC) Related to Laboratory Values
Time Frame: Baseline up to 14 days after last dose of study drug (14 days after Day 1 of Period 2 )
Population: Safety analysis set included all participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | TAK-536TCH Fasted | TAK-536TCH Fed
Number analyzed (Participants) | 12 | 12
participants | 1 | 0

15. Secondary Outcome: Number of Participants With Clinical Significant Findings in Electrocardiograms After Study Drug Administration
Description: Participants whose results of electrocardiograms were judged as abnormal and clinically significant by investigator after study drug administration were counted in this measurement.
Time Frame: Baseline up to 14 days after last dose of study drug (14 days after Day 1 of Period 2 )
Population: Safety analysis set included all participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | TAK-536TCH Fasted | TAK-536TCH Fed
Number analyzed (Participants) | 12 | 12
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 14 days for a serious adverse event after the last dose of study drug (14 days after Day 1 of Period 2).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-536TCH Fasted | TAK-536TCH Fed
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-536TCH Fasted (N=12) | TAK-536TCH Fed (N=12)
Faeces soft (Gastrointestinal disorders) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.